CLINICAL TRIAL: NCT01197287
Title: A Randomized, Double-blind, Placebo-controlled Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Doses of QAK423 in Healthy Subjects and COPD Patients and Multiple, Titrated Dosing in COPD Patients
Brief Title: Safety, Tolerability and Pharmacokinetics of QAK423A in Healthy Volunteers and Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAK423A2101
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- QAK423A Arm A (Experimental)
  Interventions: Drug: QAK423A
- QAK423A Arm B (Experimental)
  Interventions: Drug: QAK423A
- QAK423A Arm C (Experimental)
  Interventions: Drug: QAK423A

INTERVENTIONS:
Drug: QAK423A
  Arms: QAK423A Arm A
Drug: QAK423A
  Arms: QAK423A Arm B
Drug: QAK423A
  Arms: QAK423A Arm C

SUMMARY:
There are three elements to this study:

* Part A: Single dose escalation in healthy subjects. 6 dose levels of QAK423 are planned in healthy volunteers.
* Part B: Single dose escalation in patients with mild/moderate COPD. 3 dose levels of QAK423 are planned in COPD patients.
* Part C: Titrated repeat dosing for a maximum of 14 days in mild/moderate COPD patients.

Repeat dosing is planned in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Healthy, male subjects aged 18-55 years of age able to provide written informed consent prior to study participation and determined as in good health by past medical history, physical examination, ECG, laboratory tests and urinalysis.

Parts B and C:

* Male or female (post menopausal or surgically sterilized) patients with COPD, aged 40-75 years, with a smoking history of at least 10 pack years (i.e. smokers or ex-smokers).
* Diagnosis of mild or moderate COPD, according to the GOLD guidelines.
* Post-bronchodilator FEV1 at screening 50-80% of predicted.
* No COPD exacerbations within the 3 months prior to dosing, no concomitant lung disease such as asthma, requirement for long term oxygen treatment or history of lung reduction surgery.
* No medical conditions that may jeopardize the subjects participation in the study
* Weigh less than 100 kg

Exclusion Criteria:

* Use of any prescription drug or over-the-counter (OTC) medication within 2 weeks prior to dosing.
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* History of clinically significant drug allergy. A known hypersensitivity to the study drug or drugs similar to the study drug.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-05; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Adverse events associated with single doses of QAK423 in healthy subjects and mild to moderate COPD | 96 hours
Adverse events associated with repeat doses in mild to moderate COPD patients | 14 days

SECONDARY OUTCOMES:
Pharmacokinetics of single and repeat doses of QAK423 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany